CLINICAL TRIAL: NCT00326508
Title: Combination Daclizumab/Denileukin Diftitox (Ontak) Therapy for the Induction of Immune Tolerance in Non-infectious Intermediate and Posterior Uveitis
Brief Title: Combination Daclizumab/Denileukin Diftitox to Treat Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060066; 06-EI-0066
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-20

CONDITIONS: Non-infectious Intermediate and Posterior Uveitis
Keywords: T Lymphocytes; IL-2 Conjugate; CD25; T Regulatory Cells; Autoimmunity; Uveitis; Daclizumab; Denileukin Diftitox; Immune Tolerance; T Cell
MeSH Terms: conditions — Uveitis, Posterior; Autoimmune Diseases; Uveitis | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This study will determine whether treatment with a combination of the drugs daclizumab and denileukin diftitox can eliminate the need for long-term daclizumab treatment in adult patients with uveitis. Denileukin diftitox kills white blood cells called lymphocytes that cause inflammation and may be the cause of uveitis.

Patients 18 years of age and older with uveitis in one or both eyes who are on daclizumab therapy and have not had a disease flareup in 6 months may be eligible for this study. Candidates are screened with a medical history, physical examination, eye examination (including vision test, examination of the front of the eye, and pupil dilation for examination of the retina at the back of the eye), blood tests and a questionnaire about their vision and daily activities.

After screening, participants undergo the following procedures:

* Daclizumab/ denileukin diftitox treatment. Patients receive their regular dose of daclizumab intravenously (through a vein). The interval between doses is increased by 1 week after each dose. When the doses are 10 weeks apart, the daclizumab is stopped. Patients who experience a flare or uveitis are treated with intravenous denileukin diftitox and possibly local injections of steroids around the eye or increasing or adding other medicines as needed to control the uveitis.
* Fluorescein angiography to look for blood vessel abnormalities in the eyes. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina (the back portion of the eye) are taken with a special camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible abnormalities.
* Ultrasound and urine tests at enrollment and after 1 year to check kidneys, lymph nodes and pelvic area.
* Blood tests at enrollment and every 3-6 months for laboratory and immunology tests and other research tests on blood cells to examine the immune response.
* Follow-up visits approximately every 6 weeks for 2 years for repeat examinations to determine the response to treatment and drug side effects.

DETAILED DESCRIPTION:
We propose to investigate the possible efficacy of combination daclizumab and denileukin diftitox therapy to induce peripheral immune tolerance in participants presenting with non-infectious intermediate and posterior uveitis. This will be performed using a Phase I/II pilot study. Subjects whose disease is controlled on daclizumab therapy will have their daclizumab-dosing interval progressively increased by one-week increments. If and when they experience signs or symptoms of an ocular flare, they will be treated with denileukin diftitox, 24 hours after which they will receive their usual dose of daclizumab. Participants may receive up to 12 such cycles of daclizumab/denileukin diftitox therapy. When the daclizumab-dosing interval is 10 weeks long or less than 10% of their CD4 T cell CD25 is occupied by daclizumab, therapy will be discontinued. Following discontinuation of daclizumab patients will be followed for recurrence of ocular disease. Failure to reach this study point after 12 cycles or disease recurrence following discontinuation of therapy will constitute a study failure. The primary outcome will be the ability of the participant to be successfully tapered off daclizumab while their disease remains quiet (vitreous haze less than or equal to Trace) at week 104 while receiving no concomitant systemic immunosuppressive medications.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to enroll in this study, a prospective participant must satisfy the following inclusion criteria.

1. Participant is 18 years of age or older. (The vast majority of T cells are produced before adulthood and the long-term consequences of inducing immune tolerance are unknown, it would thus seem prudent to exclude juveniles from the study.)
2. Participant with uveitis in one or both eyes on daclizumab therapy without disease flare in the past 6 months.
3. Participants of reproductive age agree to use acceptable birth control methods throughout the course of the study and for 6 months after completion of treatment with daclizumab or sirolimus.
4. Participant must be willing and prepared to travel to NIH on short notice for treatment and to be hospitalized if deemed medically necessary.
5. Participant is able to understand and sign a consent form before entering the study.

EXCLUSION CRITERIA:

To be eligible to enroll in this study, a prospective participant must not satisfy any of the following exclusion criteria.

1. Participant with a history of hypersensitivity to denileukin diftitox.
2. Participant is pregnant or lactating.
3. Participant with active chronic or acute infections.
4. Participant with a history of cardiovascular disease, significant respiratory disease, coagulation disorders, or other major medical illnesses that may limit their ability to tolerate the toxicities associated with denileukin diftitox.
5. Participant with a serum albumin less than 3.0.
6. Participant with malignancy other than squamous cell carcinoma in situ.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2006-05-11; Study Completion 2006-12-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Herve P, Wijdenes J, Bergerat JP, Bordigoni P, Milpied N, Cahn JY, Clement C, Beliard R, Morel-Fourrier B, Racadot E, et al. Treatment of corticosteroid resistant acute graft-versus-host disease by in vivo administration of anti-interleukin-2 receptor monoclonal antibody (B-B10). Blood. 1990 Feb 15;75(4):1017-23. PMID 2136244